CLINICAL TRIAL: NCT05052307
Title: Effectiveness of Pfizer-BioNTech BNT162b2 mRNA COVID-19 Vaccine on Symptomatic SARS-CoV-2 Infection and COVID-19-related Hospitalizations, Mortality, and Long-term Consequences in Brazil: a Real-world Evidence Study
Brief Title: A Real-world Evidence Study of BNT162b2 mRNA Covid-19 Vaccine in Brazil
Status: Completed | Type: Observational
Sponsor: Hospital Moinhos de Vento (Other)
Collaborators: Universidade Federal do Paraná (Other); Pfizer (Industry); Inova Medical (Other)
Responsible Party: Sponsor
Other Study IDs: BNT162b2 in Toledo, Brazil
Record Dates: First submitted 2021-09-17; First posted 2021-09-22 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-02

CONDITIONS: Covid19
Keywords: COVID-19; Mass vaccination
MeSH Terms: conditions — COVID-19 | interventions — sinovac COVID-19 vaccine; Ad26COVS1

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (6):
- Fully vaccinated with BNT162b2 COVID-19 vaccine: Defined as 2 doses of Pfizer/BioNTech BNT162b2 mRNA COVID-19 vaccine received with ≥7 days between receipt of the 2nd dose and acute respiratory illness (ARI) symptom onset. This group will serve as the 'exposed' group evaluated in the primary objective.
  Interventions: Drug: Pfizer/BioNTech BNT162b2 mRNA COVID-19 vaccine
- Ever vaccinated with BNT162b2 COVID-19 vaccine: defined as ≥1 dose of Pfizer/BioNTech BNT162b2 mRNA COVID-19 vaccine received with ≥14 days between receipt of the 1st dose and ARI symptom onset.
  Interventions: Drug: Pfizer/BioNTech BNT162b2 mRNA COVID-19 vaccine
- Partially vaccinated with BNT162b2 COVID-19 vaccine: Defined as 1 dose (only) of Pfizer/BioNTech BNT162b2 mRNA COVID-19 vaccine received with ≥14 days between receipt of the 1st dose and ARI symptom onset.
  Interventions: Drug: Pfizer/BioNTech BNT162b2 mRNA COVID-19 vaccine
- Fully vaccinated with other available COVID-19 vaccines: Defined as fully vaccinated with available COVID-19 vaccines other than the BNT162b2 according to the manufacturer recommendations.
  Interventions: Drug: CoronaVac COVID-19 vaccine; Drug: ChAdOx1 nCoV-19 Covid-19 Vaccine; Drug: Ad26.COV2.S COVID-19 Vaccine
- Never vaccinated: Defined as never received any COVID-19 vaccine. This group will serve as the reference exposure group (i.e., 'unexposed' group) in all vaccine effectiveness analyses.
- Fully vaccinated plus booster dose of BNT162b2 COVID-19 vaccine: Defined as fully vaccinated with available COVID-19 vaccines according to the manufacturer recommendations plus booster dose of BNT162b2 COVID-19 vaccine received with ≥14 days between receipt of the 1st dose and ARI symptom onset.
  Interventions: Drug: Pfizer/BioNTech BNT162b2 mRNA COVID-19 vaccine; Drug: CoronaVac COVID-19 vaccine; Drug: ChAdOx1 nCoV-19 Covid-19 Vaccine; Drug: Ad26.COV2.S COVID-19 Vaccine

INTERVENTIONS:
Drug: Pfizer/BioNTech BNT162b2 mRNA COVID-19 vaccine — Pfizer/BioNTech BNT162b2 mRNA COVID-19 vaccine
  Groups: Ever vaccinated with BNT162b2 COVID-19 vaccine; Fully vaccinated plus booster dose of BNT162b2 COVID-19 vaccine; Fully vaccinated with BNT162b2 COVID-19 vaccine; Partially vaccinated with BNT162b2 COVID-19 vaccine
Drug: CoronaVac COVID-19 vaccine — CoronaVac COVID-19 vaccine
  Groups: Fully vaccinated plus booster dose of BNT162b2 COVID-19 vaccine; Fully vaccinated with other available COVID-19 vaccines
Drug: ChAdOx1 nCoV-19 Covid-19 Vaccine — ChAdOx1 nCoV-19 Covid-19 Vaccine
  Groups: Fully vaccinated plus booster dose of BNT162b2 COVID-19 vaccine; Fully vaccinated with other available COVID-19 vaccines
Drug: Ad26.COV2.S COVID-19 Vaccine — Ad26.COV2.S COVID-19 Vaccine
  Groups: Fully vaccinated plus booster dose of BNT162b2 COVID-19 vaccine; Fully vaccinated with other available COVID-19 vaccines

SUMMARY:
The present test-negative design study aims to estimate the real-world effectiveness of Pfizer-BioNTech BNT162b2 mRNA vaccine on symptomatic SARS-CoV-2 infection and its consequences following a mass vaccination campaign in the city of Toledo in Southern Brazil.

Individuals aged 12 years or older who seek the public healthcare system with symptoms suggestive COVID-19 will be enrolled. Participants with a positive polymerase chain reaction (PCR) test for SARS-CoV-2 will be classified as cases, and those with negative PCR test for SARS-CoV-2 will be classified as controls. Cases will be followed-up for a period of one year by means of structured telephone interviews.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 12 years old;
* Resident of Toledo city;
* Seeking care in the public healthcare system with symptoms suggestive of COVID-19 defined as follows: 1) ARI symptoms (nasal congestion, rhinorrhea, anosmia, sore throat, hoarseness, new or increased-from-baseline cough, sputum production, dyspnea, wheezing, myalgia) OR 2) Admitting diagnosis suggestive of ARI (pneumonia, upper respiratory infection, bronchitis, influenza, cough, asthma, viral respiratory illness, respiratory distress, AND/OR respiratory failure).
* Nasal sample for SARS-CoV-2 diagnosis obtained as standard of care.

Exclusion Criteria:

* SARS-CoV-2-directed antiviral treatment within the past 30 days;
* COVID-19 monoclonal antibody therapy within the past 90 days;
* COVID-19 convalescent serum therapy within the past 90 days;
* Lack of consent to participate.

Min Age: 12 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The present study population will be composed by individuals aged 12 years or older who seek the public healthcare system of Toledo city with symptoms suggestive COVID-19. Participants with a positive polymerase chain reaction (PCR) test for SARS-CoV-2 will be classified as cases, and those with negative PCR test for SARS-CoV-2 will be classified as controls.
Sampling Method: Non-Probability Sample
Enrollment: 4574 (Actual)
Dates: Start 2021-11-03 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2023-07-20 (Actual)

PRIMARY OUTCOMES:
Odds of symptomatic SARS-CoV-2 infection | At the moment of enrollment
  Odds of symptomatic SARS-CoV-2 infection defined by the presence of symptoms suggestive COVID-19 with a positive PCR test for SARS-CoV-2. Symptoms suggestive of COVID-19 are defined as follows: 1) Acute respiratory illness symptoms (nasal congestion, rhinorrhea, anosmia, sore throat, hoarseness, new or increased-from-baseline cough, sputum production, dyspnea, wheezing, myalgia) OR 2) Admitting diagnosis suggestive of ARI (pneumonia, upper respiratory infection, bronchitis, influenza, cough, asthma, viral respiratory illness, respiratory distress, AND/OR respiratory failure).

SECONDARY OUTCOMES:
Odds of symptomatic SARS-CoV-2 infection due to Gamma variant | At the moment of enrollment
  Odds of symptomatic SARS-CoV-2 infection due to Gamma variant defined by the presence of symptoms suggestive COVID-19 with a positive PCR test for SARS-CoV-2 Gamma variant
Odds of symptomatic SARS-CoV-2 infection due to other circulating variants of concern | At the moment of enrollment
  Odds of symptomatic SARS-CoV-2 infection due to other circulating variants of concern defined by the presence of symptoms suggestive COVID-19 with a positive PCR test for SARS-CoV-2 Alfa, Beta, or Delta variant
Duration of COVID-19 symptoms | within 180 days from enrollment
  Length of COVID-19-related symptoms
Incidence of hospitalization due to COVID-19 | Within 30 days from enrollment
  Incidence of hospital admission due to COVID-19
Incidence of ICU admission | Within 30 days from enrollment
  Incidence of ICU admission
Incidence of mechanical ventilation | Within 30 days from enrollment
  Incidence of invasive mechanical ventilation
Mortality due to COVID-19 | Within 90 days from enrollment
  Incidence of COVID-19-related mortality
Utility score of health-related quality of life at 3 months | 90 days after enrollment
  Utility score of health-related quality of life assessed with the EuroQol- 5 dimensions 3-level questionnaire. The utility score derived from the descriptive system for the Brazilian population ranges from -0.176 (indicating the worst health status [serious problems in all domains]) to 1.0 (indicating the best health status [no problems at all])
Prevalence of long COVID-19 symptoms at 6 months | 180 days after enrollment
  Incidence of long COVID-19-related symptoms (fatigue, muscular weakness, dyspnea, cough, loss of taste or smell, concentration or memory difficulties, sleep disorders, headache, anxiety, and depression)
Incidence of new symptomatic COVID-19 infection | 365 days from enrollment
  Incidence of new symptomatic COVID-19 infection defined as recurrence of COVID-19-related symptoms with a positive PCR test for SARS-CoV-2 90 days after the index infection
Incidence of any vaccine-related adverse event | 365 days from enrollment
  Incidence of any vaccine-related adverse event including local pain, hyperemia or necrosis; fever; fatigue; headache; myalgia; arthralgia; vomiting; diarrhea; and other symptoms
Incidence of vaccine-related severe adverse event | 365 days from enrollment
  Incidence of any adverse event that result in death, hospitalization or prolongation of hospitalization, and persistent or significant disability

CONTACTS AND LOCATIONS:
Overall Officials: Regis G Rosa, MD, PhD, Principal Investigator — Hospital Moinhos de Vento; Maicon Falavigna, MD, PhD, Principal Investigator — Hospital Moinhos de Vento
Locations (3):
- Brazil (3):
  - Pronto Atendimento Municipal de Toledo, Toledo, Paraná
  - Unidade Básica de Saúde Jardim Cosmos, Toledo, Paraná
  - Unidade de Pronto Atendimento Pediátrico Dr. José Ivo Alves da Rocha, Toledo, Paraná

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goulart Rosa R, Spinardi J, Allen KE, Manfio J, de Araujo CLP, Cohen M, Robinson CC, Sganzerla D, Ferreira D, de Souza EM, de Oliveira JC, Gradia DF, Brandalize APC, Kucharski GA, Pedrotti F, Rodrigues CO, Kyaw MH, Castillo GDCM, Srivastava A, McLaughlin JM, Falavigna M. BNT162b2 against COVID-19 in Brazil using a test-negative design: Study protocol and statistical analysis plan. PLoS One. 2022 Oct 20;17(10):e0276384. doi: 10.1371/journal.pone.0276384. eCollection 2022. PMID 36264905
- [Background] Rosa RG, Falavigna M, Manfio JL, de Araujo CLP, Cohen M, do Valle Barbosa GRG, de Souza AP, Romeiro Silva FK, Sganzerla D, da Silva MMD, Ferreira D, de Oliveira Rodrigues C, de Souza EM, de Oliveira JC, Gradia DF, Brandalize APC, Royer CA, Luiz RM, Kucharski GA, Pedrotti F, Valluri SR, Srivastava A, Juliao VW, Melone OC, Allen KE, Kyaw MH, Spinardi J, Del Carmen Morales Castillo G, McLaughlin JM; Toledo BNT16b2 Study Group Investigators. BNT162b2 mRNA COVID-19 against symptomatic Omicron infection following a mass vaccination campaign in southern Brazil: A prospective test-negative design study. Vaccine. 2023 Aug 23;41(37):5461-5468. doi: 10.1016/j.vaccine.2023.07.038. Epub 2023 Jul 26. PMID 37507274